CLINICAL TRIAL: NCT01826669
Title: Chest Wall Muscle Stretching and Acute Effects on Volume Variation of Thoracoabdominal Wall and Electromyographic Activity in Chronic Obstructive Pulmonary Disease
Brief Title: Chest Wall Muscle Stretching and Acute Effects in Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Rafaela Barros de Sa, Principal Investigator, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 007
Record Dates: First submitted 2012-09-14; First posted 2013-04-08 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stretching (Active Comparator): The respiratory muscle stretching were developed bilaterally as follows:
  * Upper trapezius: head lateral flexion with a hand therapist supports the the occipital region and his shoulder, promotes the stretching;
  * Sternocleidomastoid: was stretched with flexion lateral and rotation of the head to the side which hands on the occipital region and in the sternal region;
  * Scalene: with one hand on the occipital region and the other in the sternum, the two points was stretched;
  * Pectoralis major: the arm was abducted, flexed the forearm and hand was in the occipital region the therapist hands in the arm and in the side of the upper chest, which was stretched craniocaudal direction;
  * Intercostal: therapist performs with both hands to mobilize and stretch the ribs in cranial-caudal directions.
  Interventions: Procedure: Stretching
- Rest (No Intervention): COPD patients were not submitted to any intervention, remaining at rest in the same place, position and time period to the treatment group.

INTERVENTIONS:
Procedure: Stretching — Patients submitted to respiratory muscle stretching related to the increase thoracic mobility. Stretching were performed in the upper trapezius, scalenes, sternocleidomastoids, major pectoral and intercostals. The muscle stretching were performed passively by a single therapist trained and experienced. The subjects were positioned supine or lateral, knees flexed in order to correct the lumbar curve. Stretching occurred during the expiratory phase, leading to muscle maximum length, with two series of ten consecutive incursions for each muscle, with an interval of one minute between series. The patients were properly informed to perform slow exhalations and pursed-lip during stretching.
  Arms: Stretching

SUMMARY:
The study hypothesis is chest wall muscle stretching increase distribution of volume variation of thoracoabdominal wall and reduce electromyographic activity of respiratory muscles in patients with Chronic Obstructive Pulmonary Disease.

DETAILED DESCRIPTION:
Randomized controlled trial involving patients with Chronic Obstructive Pulmonary Disease evaluated before and immediately after a program of stretching muscles of the rib cage or after resting with time similar to the intervention, as volume variation of thoracoabdominal wall by optoelectronic plethysmography and on the electromyographic activity of accessory muscles of respiration.

ELIGIBILITY:
Inclusion Criteria:

* clinical and functional diagnosis of Chronic obstructive pulmonary disease according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD, 2009),
* forced expiratory volume in one second (FEV1) less than 80% predicted post-bronchodilator;
* clinical stability during the study,
* both sexes,
* age above 40 years,
* body mass index (BMI) between 18.5 and 29.9 kg / m²;
* smoking history,
* symptoms of cough,
* dyspnea or hypersecretion,
* ex-smokers for at least three months.

Exclusion Criteria:

* Disease exacerbation for at least eight weeks,
* patients with other respiratory diseases,
* cardiovascular or osteoarticular and
* participants in pulmonary rehabilitation programs.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-05; Primary Completion 2011-05 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Distribution of volume variation of thoracoabdominal wall and electromyographic activity of respiratory muscles | 1 hour

SECONDARY OUTCOMES:
Respiratory rate, minute volume, expiratory time, inspiratory time, relation inspiratory time/ total time | 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- UFPE, Recife, Pernambuco, Brazil